CLINICAL TRIAL: NCT01288729
Title: Duration of Infusion Set Function: A Study Comparing the Quick-Set Teflon Catheter vs Sure-T Steel Infusion Set Catheter
Brief Title: Duration of Infusion Set Function: Quick-Set Teflon Catheter Versus Sure-T Steel Infusion Set Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Bruce A. Buckingham, Principle Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SU-01272011-7439
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - Steel Cathetar, then Teflon (Experimental): Participants will alternate between wearing the Sure-T Steel Infusion Set Catheter for 7 days, then the Quick-Set Teflon for 7 days.They will wear each set twice starting with the Sure-T Steel Infusion Set.
  Interventions: Device: Sure-T Steel Infusion Set Catheter; Device: Quick-Set Teflon Catheter
- Group 2 - Teflon Cathetar, the Steel (Experimental): Participants will alternate between wearing the Quick-Set Teflon catheter for 7 days, then the Quick-Set Teflon for 7 days. They will wear each set twice starting with the Quick-Set Teflon set.
  Interventions: Device: Sure-T Steel Infusion Set Catheter; Device: Quick-Set Teflon Catheter

INTERVENTIONS:
Device: Sure-T Steel Infusion Set Catheter — Participants will wear Quick-Set Teflon Catheter or Sure-T Steel Infusion Set Catheter for 2 weeks each during the active study time
Device: Quick-Set Teflon Catheter — Participants will wear Quick-Set Teflon Catheter or Sure-T Steel Infusion Set Catheter for 2 weeks each during the active study time

SUMMARY:
This is an open-label cross over study looking to compare the length of infusion set wear between a teflon catheter (Quick-Set) or a steel (Sure-T) catheter.

DETAILED DESCRIPTION:
Currently infusion sets are approved for 2-3 days of wear. In this study subjects will wear each infusion set for up to 7 days or until the infusion set fails. Subjects will alternate between wearing the Quick-Set Teflon catheter and the Sure-T steel catheter each week. They will wear each infusion set twice.

For the study, subjects will be provided with an investigational Medtronic Real-Time Continuous Glucose Monitor (CGM) Enlite Sensor/Serter to help identify, serious hyperglycemia or hypoglycemia during the study. This sensor is not yet FDA approved, but is similar to commercially available sensors. If the sensor detects a high or low glucose, subject must obtain a fingerstick glucose to confirm the result. In the study, all insulin dose and other treatment decisions will be made using glucose meter results, and will not be based on sensor results. Subjects will be instructed on how to identify infusion set failures.

Infusion set failure are defined as: 1) Blood ketones greater than 0.6 mmol/L, 2) Evidence of infection at the infusion site (such as redness of more than 4 mm), or 3) Blood glucose that does not decrease by at least 50 mg/dL within 1 hour of a correction bolus to treat a blood glucose greater than 300 mg/dL.

Subjects will follow-up weekly in one of our test centers for a total of five visits.

At home subjects will be asked to keep a log recording measurements of redness and induration at the infusion site when it is changed prior to the study visit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least one year and using an insulin pump for at least 3 months
* The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
* Age 12 to 45 years
* For females, not currently known to be pregnant
* An understanding of and willingness to follow the protocol and sign the informed consent
* Hemoglobin A1c level less than or equal to 10%
* Medtronic Continuous subcutaneous insulin infusion pump
* Must be able to understand spoken or written English

Exclusion Criteria:

* Diabetic ketoacidosis in the past 6 months
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 6 months prior to enrollment
* Current treatment for a seizure disorder
* Cystic fibrosis
* Active infection
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:
* Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian)
* Presence of a known adrenal disorder
* If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
* Abuse of alcohol

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A. Buckingham, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patel PJ, Benasi K, Ferrari G, Evans MG, Shanmugham S, Wilson DM, Buckingham BA. Randomized trial of infusion set function: steel versus teflon. Diabetes Technol Ther. 2014 Jan;16(1):15-9. doi: 10.1089/dia.2013.0119. Epub 2013 Oct 3. PMID 24090124

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Steel Cathetar, Then Teflon: Participants will alternate between wearing the Sure-T Steel Infusion Set Catheter for 7 days, then the Quick-Set Teflon for 7 days.They will wear each set twice starting with the Sure-T Steel Infusion Set.
Period: Overall Study
Arm/Group | Group 1: Steel Cathetar, Then Teflon | Group 2 - Teflon Cathetar, the Steel
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Steel Cathetar, Then Teflon | Group 2 - Teflon Cathetar, the Steel | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (8.8) | 22.3 (8.8) | 22.3 (8.8)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Length of Wear of Infusion Site
Description: Comparison of the length of wear (hours) of Sure-T Steel Infusion Set Catheter versus Quick-Set Teflon Catheter. Infusion sets are currently approved for wear 2-3 days (24-72 hours). Participants wore each set for up to 7 days twice. Outcome measure is presented according to the intervention (Steel or Teflon catheter).
Time Frame: 5 weeks
Population: Participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Sure-T Steel Infusion Set Catheter: Participants will wear Sure-T Steel Infusion Set Catheter for 7 days (for a total of 14 days for the duration of the study)
  Sure-T Stell Infusion Set Catheter: Participants will wear Quick-Set Teflon Catheter or Sure-T Steel Infusion Set Catheter for 2 weeks each during the active study time
  Quick-Set Teflon Catheter: Participants will wear Quick-Set Teflon Catheter or Sure-T Steel Infusion Set Catheter for 2 weeks each during the active study time
- Quick-Set Teflon Catheter: Participants will wear the Quick-Set Teflon catheter for 7 days (for a total of 14 days for the duration of the study).
  Sure-T Stell Infusion Set Catheter: Participants will wear Quick-Set Teflon Catheter or Sure-T Steel Infusion Set Catheter for 2 weeks each during the active study time
  Quick-Set Teflon Catheter: Participants will wear Quick-Set Teflon Catheter or Sure-T Steel Infusion Set Catheter for 2 weeks each during the active study time
Arm/Group | Sure-T Steel Infusion Set Catheter | Quick-Set Teflon Catheter
Number analyzed (Participants) | 19 | 20
hours | 137 [87 to 168] | 145 [99 to 167]

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: Safety data is presented according to the intervention (Steel or Teflon catheter).
Arm/Group | Sure-T Steel Infusion Set Catheter | Quick-Set Teflon Catheter
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 7/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sure-T Steel Infusion Set Catheter (N=20) | Quick-Set Teflon Catheter (N=20)
Skin reaction to infusion set (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) — redness and/or induration
ketosis (Endocrine disorders) | 2 (2) | 4 (4) — serum ketones >0.6 mmol/L

LIMITATIONS AND CAVEATS:
This was a single center study with 20 subjects enrolled in a cross-over study. A larger study would make results more robust. In addition, if each subject had worn each infusion set 3 to 6 times, it would make the study more robust.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No